CLINICAL TRIAL: NCT02344693
Title: Electroencephalography in Patients Resuscitated From Cardiac Arrest
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Johannes Björkman, Resident, Helsinki University Central Hospital
Other Study IDs: 237/4 03.12.2012
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Cardiac Arrest; Heart Arrest
Keywords: Electroencephalography
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Sudden cardiac death can occur due to a multitude of causes. The underlying case can affect the overall prognosis. A return of spontaneous circulation not exceeding 30 minutes following a successful cardiopulmonary resuscitation is usually deemed imperative, if the patient is to survive. Monitors for evaluating the cardiac function during and after resuscitation are implemented on a daily basis (ekg, pulseoxymetry, blood pressure monitoring, cardiac sonography), but no devices for registration of the cortical brain activity exist. The aim of this study is to provide a 3-channel electroencephalogram using a prototype EEG/EKG adapter, connected to a Physio-Control LifePak 15 monitor/defibrillator, in patients who regain spontaneous circulation following non-traumatic cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed Cardiac Arrest
* Return of spontaneous circulation following cardiac arrest 10-40 min

Exclusion Criteria:

* traumatic cardiac arrest
* no consent from next-of-kin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients resuscitated from a non-traumatic cardiac arrest in a urban setting in southern Finland
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
prehospital EEG value in regard to patient discharge | 60-min

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Björkman, MD, Principal Investigator — Helsinki University Central Hospital; Tom Silfvast, MD, PhD, Study Director — Helsinki University Central Hospital; Tapani Salmi, MD, PhD, Study Director — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland